CLINICAL TRIAL: NCT02343809
Title: Effectiveness of Diacutaneous Fibrolysis on Chronic Lateral Epicondylitis. A Randomized Controlled Trial.
Brief Title: Diacutaneous Fibrolysis on Lateral Epicondylitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P14/032
Record Dates: First submitted 2015-01-16; First posted 2015-01-22 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Tennis Elbow
Keywords: Physiotherapy; Lateral epicondylitis; Manual therapy
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Intervention Group (Experimental): Actual Diacutaneous Fibrolysis and Protocolized Physiotherapy
  Interventions: Other: Actual Diacutaneous Fibrolysis; Other: Protocolized Physiotherapy
- Placebo Group (Sham Comparator): Sham Diacutaneous Fibrolysis and Protocolized Physiotherapy
  Interventions: Other: Sham Diacutaneous Fibrolysis; Other: Protocolized Physiotherapy
- Control Group (Other): Protocolized Physiotherapy
  Interventions: Other: Protocolized Physiotherapy

INTERVENTIONS:
Other: Actual Diacutaneous Fibrolysis — Diacutaneous Fibrolysis is a non-invasive physiotherapeutic technique applied by means of a set of metallic hooks ending in a spatula with bevelled edges that allow a deeper and more precise application, which could not be achieved manually. The hook is deeply applied following the intermuscular septum between the muscles with an anatomical of functional relationship with the painful structure in order to release adherences between musculoskeletal structures.
  Arms: Intervention Group
Other: Sham Diacutaneous Fibrolysis — Sham Diacutaneous Fibrolysis is applied at a superficial level. A pinch of skin was held with the thumb of the palpatory hand and the tip of the spatula, without any action taking place on the deep tissular levels.
  Arms: Placebo Group
Other: Protocolized Physiotherapy — Protocolized physiotherapeutic treatment: Three weeks fo daily stretching exercises, ultrasound and analgesic electrotherapy

SUMMARY:
Diacutaneous Fibrolysis (DF) is a manual method of treatment, usually adjuvant, addressed to the mechanical pain of the locomotor system. In our clinical practice a favorable effect is observed in patients with chronic lateral epicondylitis, but there are no published studies evaluating the results of this technique.

The objective of this trial is to evaluate if DF provides a further improvement in pain intensity, pain-pressure threshold, function and pain-free grip strength, in patients with chronic lateral epicondylitis being treated with physiotherapy. For this purpose, we conduct a randomized controlled trial, double-blind (patient and evaluator) in a Public Primary Care Center.

Sixty subjects will be randomized (computer application) into three groups: Intervention Group, Placebo Group and Control Group. All the three groups receive the same protocolized treatment of physiotherapy and additionally. Additionally, the Intervention Group receives six sessions (two sessions in a week during three weeks) of real DF and the Placebo Group receives six sessions (two sessions in a week during three weeks) of sham DF. The Control Group receives the protocolized treatment of physiotherapy only.

Pain intensity (VAS), pain-pressure threshold (pressure algometry), function (DASH questionnaire) and pain-free grip strength (digital dynamometer) will be measured at baseline, after treatment period, and three months after discharge from treatment. After discharge for treatment the patient subjective opinion about their evolution will be collected through the Global Rating of Change (GROC) scale.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and over
* Diagnosis of chronic lateral epicondylalgia
* Sign the informed consent form

Exclusion Criteria:

* Concomitant conditions affecting the same upper extremity
* Contraindications for Diacutaneous Fibrolysis
* Corticosteroid injections or similar agents in the three months prior to study inclusion
* Pending litigation or legal claim
* Poor language and communication skills making difficult to understand the informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-10; Primary Completion 2015-11 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | pre-intervention, post-intervention (two sessions in a week during three weeks), after three months
  Pain intensity (VAS)

SECONDARY OUTCOMES:
Pressure Pain Threshold | pre-intervention, post-intervention (two sessions in a week during three weeks), after three months
  pressure algometry
Pain free grip strength | pre-intervention, post-intervention (two sessions in a week during three weeks), after three months
  digital dynamometer
Functional status | pre-intervention, post-intervention (two sessions in a week during three weeks), after three months
  DASH questionnaire
Global Rating of Change scale | post-intervention, after three months

CONTACTS AND LOCATIONS:
Locations (1):
- Catalan Institut of Health - Sant Ildefons Rehabilitation Center, Cornellà de Llobregat, Barcelona, Spain